CLINICAL TRIAL: NCT05588557
Title: A Phase I Dose-escalation Study, Randomized Comparison with Active Control to Evaluate the Safety and Pharmacokinetics of a Single Administration of ND-340 Via Adductor Canal Block (ACB) and IPACK Block in Healthy Volunteers
Brief Title: A Phase I Study to Evaluate the Safety and PK of ND-340 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nang Kuang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKC340-202101
Record Dates: First submitted 2022-07-04; First posted 2022-10-20 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Pain, Postoperative
Keywords: Bupivacaine; Pharmacokinetics; Analgesics
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Injections

STUDY DESIGN:
Intervention Model Description: The subjects of each cohort will be randomly arranged to receive ND-340 or control drug (Marcaine® Injection 0.5%, equal to bupivacaine base 5 mg/mL) in the ratio of 3:1.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Marcaine® 100mg/20mL (0.5%) bupivacaine solution for Injection (Active Comparator): Marcaine® at 150 mg in each cohort.
  Interventions: Drug: Marcaine® 100mg/20mL (0.5%) bupivacaine solution for Injection
- ND-340 (Bupivacaine Microsphere), 300 mg/vial bupivacaine for extended-release injectable suspension (Experimental): ND-340(90-320 mg) at dose escalations
  Interventions: Drug: ND-340 (Bupivacaine Microsphere), 300 mg/vial bupivacaine for extended-release injectable suspension

INTERVENTIONS:
Drug: Marcaine® 100mg/20mL (0.5%) bupivacaine solution for Injection — Subjects in this arm will receive a single administration of Marcaine® at the 150 mg.
  Marcaine® will be administered under ultrasound guidance with a total volume of 40 mL, of which 20 mL will be used via adductor canal block (ACB) and the other 20 mL will be used as IPACK block (interspace between the popliteal artery and the capsule of the posterior knee).
  Arms: Marcaine® 100mg/20mL (0.5%) bupivacaine solution for Injection
Drug: ND-340 (Bupivacaine Microsphere), 300 mg/vial bupivacaine for extended-release injectable suspension — Subjects in this arm will receive a single administration of ND-340 at the specified dose (90-320 mg).
  ND-340 will be administered under ultrasound guidance with a total volume of 40 mL, of which 20 mL will be used via adductor canal block (ACB) and the other 20 mL will be used as IPACK block (interspace between the popliteal artery and the capsule of the posterior knee).
  Arms: ND-340 (Bupivacaine Microsphere), 300 mg/vial bupivacaine for extended-release injectable suspension

SUMMARY:
This study focuses on ND-340 extended release injection suspension for healthy volunteers with a one-time nerve blockade to determine the safety, tolerability, and pharmacokinetic profile.

DETAILED DESCRIPTION:
The current investigational product, ND-340, is a bupivacaine microsphere injection with an extended release profiling. Lipid microsphere, or liposphere, has been proposed as new type of lipid-based encapsulation system for drug delivery of bioactive compounds especially lipophilic compound.

ND-340 has not been studied in human before. However, MARCAINE® and EXPAREL® are both FDA-approved drugs, which contain the same active pharmaceutical ingredient (API) as ND-340, which is bupivacaine. MARCAINE® is indicated for the production of local or regional anesthesia or analgesia for surgery, dental and oral surgery procedures, diagnostic and therapeutic procedures, and for obstetrical procedures.

In this study, Investigators will focus on determining the safety, tolerability, and pharmacokinetic profile of ND-340.

ELIGIBILITY:
Inclusion Criteria:

1. 20 - 45 year-old healthy male subjects or female subjects who are in non-lactating and non-pregnant status.
2. Subjects must have a Body Mass Index (BMI) of 18.5 to 30.0 Kg/m², inclusive. For male subjects, body weight must be above 50 kg; for female subjects, body weight must be above 45 kg. BMI = Weight (kg)/Height (m2).
3. Female subject with childbearing potential must have a negative serum pregnancy test at the screening visit.
4. Able and willing to comply with all study visits and procedures.
5. The informed consent form has been read, signed and dated by the subject.
6. Able to communicate well with the investigator, comply with study questionnaires, and other instruments used for collecting subject-reported outcomes.

Exclusion Criteria:

1. Subject has a sitting pulse rate outside the reference range of 50 to 90 beats per minute or an ear temperature outside the reference range of 35.0 to 37.5°C or a sitting blood pressure less than 90/50 mmHg or more than 140/90 mmHg at screening visit.
2. Subject has clinically significant results of physical examination, laboratory tests, electrocardiogram, or chest X-ray as judged by the investigator at the screening visit.
3. With abnormal results of sensory and neurological assessment as judged by the investigator at the screening visit.
4. Presence of liver disease or liver injury as indicated by an abnormal liver function profile such as alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkalinephosphatase (ALP), or total bilirubin, if any one of them is out of the reference range.
5. Presence of impaired renal function as indicated by abnormal creatinine or blood urea nitrogen values or abnormal urinary constituents, if any one of them is out of the reference range.
6. Known of active infection with HIV, HBV, or HCV as defined by blood tests at the screening visit.
7. Presence of clinically significant illness, such as cardiovascular disease, cerebrovascular disease, metabolic disease, respiratory disease, neurological disease, psychiatric disease, cancers or immunological disease, may increase the risk of study as judged by the investigator at the screening visit.
8. Subject does not agree not to take any prescription, over-the-counter medication, herbal medicine and dietary supplement (including multivitamins) within two weeks before hospital admission and until the end of the study.
9. Subject does not agree not to consume any beverage or food that might affect the drug metabolism, such as pomelo, grapefruit or related products within one week before hospital admission and until the end of the study.
10. Subject does not agree not to consume any caffeine-containing product (e.g., tea, coffee, coke, or chocolate) 3 days prior to hospital admission and until the end of the study.
11. Subject does not agree not to consume any product containing tobacco, nicotine (such as e-cigarettes, nicotine gum), and alcohol 3 days prior to hospital admission and until the end of the study.
12. Administration of an investigational drug within 2 months or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration; or planned administration of another investigational product or procedure during the study period.
13. Donation or loss of more than 500 mL and 250 mL of blood within 3 months and 2 months before the screening visit, respectively.
14. Known with a history of allergy or hypersensitivity to medicine as judged by the investigator at the screening visit.
15. Female subject who is breast-feeding, pregnant, or planning to become pregnant.
16. Subject does not agree to use effective non-hormonal contraception method to prevent from pregnancy ('double barrier method': condoms used concomitantly with vaginal sponge, diaphragm or intra-uterine contraceptive device) or abstain from sexual behavior with his/her partner from screening until the end of the study.
17. Individual is not eligible to be a subject for other reasons based on the judgment of investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Adverse events as assessed by CTCAE v 5.0 | From administration of ND-340 to 140 hours
  Treatment-related adverse events will be analyzed by cohort
Changes in 12-lead ECG and Holter monitor | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hour
  To definition safety profile in cardiac events, vent. rate, PR interval, QRS duration, QT interval, QTc interval
Changes in Laboratory test - hematology | Pre-dose, 140 hour
  Hemoglobin, Hct, RBC count, WBC count, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, Platelet count
Changes in Laboratory tests - biochemistry | Pre-dose, 140 hour
  Albumin, Total protein, ALT, AST, ALP, Total bilirubin, BUN, Serum creatinine, K, Na, Mg, Ca, P, Uric acid, Total cholesterol, HbA1c
Changes in Laboratory tests - urinalysis | Pre-dose, 140 hour
  pH, Specific gravity, Leukocyte, Erythrocyte, Protein, Glucose
Changes in vital signs | Screening visit, day 0 (Pre-dose, 60 mins), Day 1, Day 2, Day 3, Day 4, Day 5, Day 6
  To definition safety profile including body temperature,blood pressure, respiratory rate, pulse rate
Changes in physical examination | Screening visit, day -1, Day 6
  To definition safety profile including general appearance, HEENT, neck, Lymph nodes, skin, cardiovascular, pulmonary, abdomen, neurological system, musculoskeletal/joints
The tolerability and maximal tolerated dose (MTD) of ND-340 by dose-limiting toxicities (DLTs) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hour
  The incidence of DLT will be summarized by each cohort. The number of subject who has DLT will be summarized by cohorts.
  and the determination of MTD in this study will be provided.
Cmax | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hours
  Maximum Plasma Concentration of ND-340
Tmax | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hours
  Time of peak concentration of ND-340
AUC 0-t | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hours
  Area under the plasma concentration versus time curve from zero to t of ND-340
AUC 0-∞ | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hours
  Area under the plasma concentration versus time curve from zero to infinity of ND-340
T1/2 | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hours
  Terminal half life of ND-340
CL/F | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hours
  Clearance/Bioavailability of ND-340
λz | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hours
  Terminal elimination rate constant
Vz/F | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hours
  Apparent volume of distribution during terminal phase after non-intravenous administration
MRT 0-∞ | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hours
  Mean residence time from zero to infinity of ND-340

SECONDARY OUTCOMES:
Range of motion of knee | Pre-dose, 1, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140 hours
  The range of motion (ROM) of knee as measured by knee flexion and extension at baseline and subsequent visits, and the change from baseline will be summarized descriptively by cohorts and drugs(ND-340 or Marcaine®).
The ambulation distance | Once a day on Pre-dose, Day 1 and Day 2
  The ambulation distance as measured by six-minute walk test (6MWT) at baseline and subsequent visits, and the change from baseline will be summarized descriptively by cohorts and drugs (ND-340 or Marcaine®).

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Peng Lin, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan